CLINICAL TRIAL: NCT03271892
Title: Deciding on Active Surveillance as an Alternative Option to Surgery in the Primary Management of Low Risk Papillary Thyroid Cancer
Brief Title: Deciding on Active Surveillance or Surgery for Primary Management of Low Risk Papillary Thyroid Cancer
Acronym: AS-PTC
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Ontario Ministry of Health and Long Term Care (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 15-8942
Record Dates: First submitted 2017-08-28; First posted 2017-09-05 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Cancer Stage I
Keywords: papillary thyroid cancer; thyroidectomy; active surveillance
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active surveillance: Patients under active surveillance choose to not have immediate thyroidectomy. Patients are closely monitored with respect to clinical status, ultrasound imaging, biochemical indices (thyroid function, thyroglobulin, and thyroglobulin antibodies) and any thyroid cancer-related treatments (if needed). Active surveillance is conducted at a participating study site. Criteria defining disease progression are established, and if such criteria are met, thyroid surgery is recommended to the patient. However, patients are free to choose to have thyroid surgery at any time, in the absence of disease progression. Thyroid cancer clinical and treatment outcomes are tracked by the study team.
- Immediate Surgery: Patients who choose surgery, undergo thyroidectomy, as per current standards of care, by a surgeon of their choice in an institution of their choice. The treating surgeon, in discussion with the patient, will choose the extent of thyroid surgery that may be appropriate for the individual case. Post-surgical follow-up is per the discretion of the treating surgeon, endocrinologist, or other healthcare providers involved in the patient's thyroid cancer care. Thyroid cancer clinical and treatment outcomes are tracked by the study team.

SUMMARY:
This is a prospective observational study.

1. In the first part of the study, consenting eligible adult patients with low risk papillary thyroid cancer that is confined to the thyroid, are provided verbal and written information about their disease and the option of active surveillance (close monitoring with intention to treat if disease progresses or if the patient changes her/his mind), as an alternative to thyroid surgery (thyroidectomy - traditional standard of care). Patients are free to make their own disease management choice (ie. active surveillance or thyroidectomy) and the investigators are examining how often patients choose each of these options. The investigators are also examining the reasons for their choice.
2. In the second part of the study, consenting, eligible patients who completed the preceding part of the study and chose either a) active surveillance, or b) thyroid surgery, are tracked with respect to clinical and psychosocial outcomes as well as quality of life. Patients who chose active surveillance are free to change their mind and have surgery at any point, even if the disease does not progress. The primary study outcome is decision regret at one year, in the respective groups of patients who chose active surveillance or thyroidectomy.

DETAILED DESCRIPTION:
This is a prospective observational study, consisting of multiple parts.

1. In the first part of the study, eligible, consenting adult patients with low risk papillary thyroid cancer who have not had thyroid surgery, are provided with verbal and written information about the disease prognosis, surgical treatment outcomes, and the option of active surveillance (close monitoring with the intention of treatment if there is disease progression or if the patient changes her/his mind), as an alternative to immediately proceeding with thyroidectomy. The primary outcome of this part of the study is the final disease management decision of the patient (ie. active surveillance or thyroid surgery) and we are also examining patients' reasons for their choice.
2. In the second part of this study, eligible consenting patients who completed the preceding part of the study and chose either: a) active surveillance, or b) thyroid surgery, are tracked with respect to disease, treatment, psychosocial outcomes, and quality of life. For patients under active surveillance, clinical follow-up is conducted at a participating study institution. For patients who choose surgery, surgery and related clinical follow-up may be performed at any institution (of the patient's choice), however, the thyroid cancer-related medical records are regularly reviewed. Questionnaires are mailed to patients at one year. The primary outcome for this study is decision regret (on the decision for active surveillance or surgery) at one year after initiating the disease management decision (ie. active surveillance or surgery). As the decision for surgery or active surveillance is up to the patient and the proportion of patients in each group is unknown, the results in respective groups will be reported separately for the primary analysis (and only compared if sufficient numbers are available in each group).

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Newly diagnosed previously untreated papillary thyroid cancer (PTC) (fine needle aspiration biopsy positive for PTC or suspicious for PTC).
3. PTC must be less than 2 cm in maximal diameter on thyroid ultrasound
4. No evidence of metastatic cervical lymphadenopathy on ultrasound imaging of the neck (or other neck imaging) and no known distant metastatic thyroid cancer.
5. No other absolute indications for thyroid or parathyroid surgery
6. Permission for review of thyroid cancer-related medical records

Exclusion Criteria:

1. Regional or distant metastatic thyroid cancer
2. History of prior thyroid cancer surgery
3. High risk location of the PTC (e.g. adjacent to the recurrent laryngeal nerve or trachea)
4. The patient has clinical signs, imaging, or indirect laryngoscopy findings suggestive of locally advanced thyroid cancer (i.e. vocal cord paralysis or any clinical or radiographic signs of extrathyroidal invasion into adjacent structures such as the strap muscles of the neck, trachea or esophagus)
5. Known or suspected poorly differentiated or non-papillary thyroid cancer
6. Medically unfit for surgery due to co-morbidity
7. Another active malignancy with limited life expectancy of < 1 year.
8. Pregnancy at the time of study enrollment.
9. Other absolute indication for thyroid or parathyroid surgery
10. Unable to provide informed consent for the study or comply with study follow-up procedures due to current severe active cognitive or psychiatric impairment, substance abuse, or other reasons.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting individuals aged 18 years of age or older with papillary thyroid cancer (PTC) who have a primary tumor that is <2cm in maximal diameter, and fine needle aspiration biopsy is positive or suspicious for PTC. The tumor must be confined to the thyroid (no metastatic disease) and not considered in a high risk location (e.g. adjacent to the recurrent laryngeal nerve or trachea). The patient must have no prior surgical treatment for thyroid cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-05-11 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease management decision (first part of the study, focused on treatment management choice) | 0 to 3 months after enrollment in the study (as it is expected that the disease management decision should be completed within that time frame)
  In the first part of the study, at any time point after study enrollment and receiving written and verbal information about disease prognosis and the option of active surveillance, patients will be asked to provide a final disease management decision (active surveillance or surgery). This decision should be generally finalized within 3 months of enrollment in the study.
Decision regret (second part of the study - follow-up of respective active surveillance and surgical patient groups) | 1 year after enrolling in the second phase of the study (i.e. one year after enrolling in the active surveillance arm or 1 year after the first thyroid cancer surgery)
  Decision regret (total score, self-administered written questionnaire)

SECONDARY OUTCOMES:
Disease management decision rationale/explanation | 0 to 3 months after enrollment in the study, once the decision on disease management is finalized (it is expected that the disease management decision should be completed within the time frame of 0 to 3 months)
  Patients will be asked the reason for choosing active surveillance or surgery once final decision is complete for the disease management plan (i.e. active surveillance or surgery). Each patient will be asked, in a semi-structured interview question, to explain the reason why the disease management strategy that was chosen. The results will be coded and analyzed using a mixed methods approach.
Disease management decision-maker identification | 0 to 3 months after enrollment in the study, once the decision on disease management is finalized (it is expected that the disease management decision should be completed within the time frame of 0 to 3 months)
  Patients will be asked about the extent of their involvement in disease management decision-making
Disease management decision satisfaction | 0 to 3 months after enrollment in the study, once the decision on disease management is finalized (it is expected that the disease management decision should be completed within the time frame of 0 to 3 months)
  Satisfaction with decision scale (overall score)
Baseline coping mechanisms in all patients and respective study groups | Within 1 month of study enrollment (baseline interview after enrollment in the study, prior to being provided detailed information about active surveillance)
  Brief Cope Questionnaire (description of all respective subscales per the questionnaire developer)
Baseline evaluation of fear of disease progression in all patients and respective study groups (i.e. those who ultimately choose active surveillance or surgery) | Within 1 month of study enrollment (baseline interview after enrollment in the study, prior to being provided detailed information about active surveillance)
  Short form of the Fear of Progression Questionnaire (overall score)
Fear of disease progression at 1 year follow-up - in respective study groups (active surveillance or surgery) | 1 year after enrolling in the second phase of the study (i.e. one year after enrolling in the active surveillance arm or 1 year after the first thyroid cancer surgery)
  Short form of the Fear of Progression Questionnaire (overall score)
Baseline evaluation of surgical fear in all patients and respective study groups (i.e. those who ultimately choose active surveillance or surgery) | Within 1 month of study enrollment (baseline interview after enrollment in the study, prior to being provided detailed information about active surveillance)
  Surgical Fear Questionnaire (total score)
Baseline evaluation of decision self-efficacy in all patients and respective study groups (i.e. those who ultimately choose active surveillance or surgery) | Within 1 month of study enrollment (baseline interview after enrollment in the study, prior to being provided detailed information about active surveillance)
  Decision Self-Efficacy Scale (total score)
Psychological distress at 1 year in respective study groups | 1 year after enrolling in the second phase of the study (i.e. one year after enrolling in the active surveillance arm or 1 year after the first thyroid cancer surgery)
  Hospital Anxiety and Depression Scale (respective total scores for anxiety and depression, respectively)
Disease-specific quality of life at 1 year | 1 year after enrolling in the second phase of the study (i.e. one year after enrolling in the active surveillance arm or 1 year after the first thyroid cancer surgery)
  M.D. Anderson Symptom Inventory (respective Symptom Severity and Symptom Interference with life - respective total scores for these subscales)
Body image perception at 1 year | 1 year after enrolling in the second phase of the study (i.e. one year after enrolling in the active surveillance arm or 1 year after the first thyroid cancer surgery)
  Body Image Scale (overall score)
Thyroid cancer surgery in patients who initially choose active surveillance | From date of enrollment in the active surveillance arm of the study until the date of first documented thyroid cancer surgery or date of death from any cause, whichever comes first, assessed up to 10 years from active surveillance arm study enrollment
  The number and percent of patients who initially choose active surveillance, but go on to have surgery (with surgical indication) will be evaluated yearly
Disease progression | From date of enrollment in the active surveillance or surgical arms of the study until the date of first documented thyroid cancer structural disease progression or death from any cause, whichever comes first, assessed up to 10 years from enrollment
  Structural disease progression (Defined as follows: primary tumor growth >3 mm in largest diameter in the active surveillance group, or new metastatic disease in either the active surveillance or surgical group, or newly diagnosed thyroid cancer in the thyroid bed/remaining thyroid lobe in the surgical group)
Thyroid surgical complications | From date of enrollment in the active surveillance or surgical arms of the study until the date of any documented thyroid cancer surgical complication or death from any cause, whichever comes first, assessed up to 10 years from enrollment
  Any thyroid surgical complications (defined as hypoparathyroidism, recurrent laryngeal nerve injury, or other surgical complications documented in the medical record) will be ascertained in all patients from either group, who undergo thyroid surgery
New chronic prescription thyroid hormone use | From date of enrollment in the active surveillance or surgical arms of the study until the date of first documented prescription thyroid hormone use or death from any cause, whichever comes first, assessed up to 10 years from enrollment
  New chronic prescription thyroid hormone use will be ascertained in both study arms. Individuals who are taking chronic prescription thyroid hormone prior to enrollment in the study will be excluded from this analysis.
Healthcare resource utilization | From the date of enrollment until death from any cause or up to 10 years from enrollment
  Thyroid cancer or thyroid cancer care-related expenses/procedures will be ascertained in both study arms including thyroid cancer surgery, thyroid hormone use, thyroid cancer-related diagnostic testing [bloodwork, imaging], thyroid biopsies, other thyroid cancer-related procedures, thyroid cancer-related specialist healthcare provider visits, radioactive iodine treatment or scans, use of recombinant human thyrotropin, or healthcare expenditures for treatments of complications of thyroid surgery [e.g. prescription treatments for hypoparathyroidism]).
Serum thyroglobulin measurement in the active surveillance group | Upon enrollment in the active surveillance arm of the study and thereafter every 6 months for 2 years, and thereafter yearly, for up to 10 years, for patients in the active surveillance arm of the study (who do not have surgery)
  Serum thyroglobulin (with thyroglobulin antibody) measurement

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Sawka, MD,PhD, Principal Investigator — University Health Network, Toronto; David P Goldstein, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We are in discussions with other groups doing active surveillance research, and in future, may share data with such groups. Final plan not yet established.

REFERENCES:
- [Background] Sawka AM, Ghai S, Rotstein L, Irish JC, Pasternak JD, Monteiro E, Chung J, Su J, Xu W, Esemezie AO, Jones JM, Gafni A, Baxter NN, Goldstein DP; Canadian Thyroid Cancer Active Surveillance Study Group (Greater Toronto Area). Long-Term Durability of Active Surveillance of Small, Low-Risk Papillary Thyroid Cancer. JAMA Surg. 2025 Oct 1;160(10):1117-1124. doi: 10.1001/jamasurg.2025.2957. PMID 40833769
- [Background] Sawka AM, Ghai S, Tomlinson G, Rotstein L, Gilbert R, Gullane P, Pasternak J, Brown D, de Almeida J, Irish J, Chepeha D, Higgins K, Monteiro E, Jones JM, Gafni A, Goldstein DP. A protocol for a Canadian prospective observational study of decision-making on active surveillance or surgery for low-risk papillary thyroid cancer. BMJ Open. 2018 Apr 12;8(4):e020298. doi: 10.1136/bmjopen-2017-020298. PMID 29654030
- [Background] Sawka AM, Ghai S, Ihekire O, Jones JM, Gafni A, Baxter NN, Goldstein DP, On Behalf Of The Canadian Thyroid Cancer Active Surveillance Study Group. Decision-making in Surgery or Active Surveillance for Low Risk Papillary Thyroid Cancer During the COVID-19 Pandemic. Cancers (Basel). 2021 Jan 20;13(3):371. doi: 10.3390/cancers13030371. PMID 33498497
- [Background] Sawka AM, Ghai S, Rotstein L, Irish JC, Pasternak JD, Gullane PJ, Monteiro E, Gooden E, Brown DH, Eskander A, Zahedi A, Chung J, Su J, Xu W, Ihekire O, Jones JM, Gafni A, Baxter NN, Goldstein DP; Canadian Active Surveillance Study Group (Greater Toronto Area). A Quantitative Analysis Examining Patients' Choice of Active Surveillance or Surgery for Managing Low-Risk Papillary Thyroid Cancer. Thyroid. 2022 Mar;32(3):255-262. doi: 10.1089/thy.2021.0485. Epub 2022 Feb 17. PMID 35019770
- [Background] Sawka AM, Ghai S, Rotstein L, Irish JC, Pasternak JD, Monteiro E, Chung J, Zahedi A, Su J, Xu W, Jones JM, Gafni A, Baxter NN, Goldstein DP. Decision Regret Following the Choice of Surgery or Active Surveillance for Small, Low-Risk Papillary Thyroid Cancer: A Prospective Cohort Study. Thyroid. 2024 May;34(5):626-634. doi: 10.1089/thy.2023.0634. Epub 2024 Apr 8. PMID 38481111
- [Background] Sawka AM, Ghai S, Rotstein L, Irish JC, Pasternak JD, Gullane PJ, Monteiro E, Zahedi A, Gooden E, Eskander A, Chung J, Devon K, Su J, Xu W, Jones JM, Gafni A, Baxter NN, Goldstein DP; Canadian Thyroid Cancer Active Surveillance Study Group (Greater Toronto Area). Gender Differences in Fears Related to Low-Risk Papillary Thyroid Cancer and Its Treatment. JAMA Otolaryngol Head Neck Surg. 2023 Sep 1;149(9):803-810. doi: 10.1001/jamaoto.2023.1642. PMID 37410454
- [Background] Sawka AM, Ghai S, Yoannidis T, Rotstein L, Gullane PJ, Gilbert RW, Pasternak JD, Brown DH, Eskander A, Almeida JR, Irish JC, Higgins K, Enepekides DJ, Monteiro E, Banerjee A, Shah M, Gooden E, Zahedi A, Korman M, Ezzat S, Jones JM, Rac VE, Tomlinson G, Stanimirovic A, Gafni A, Baxter NN, Goldstein DP. A Prospective Mixed-Methods Study of Decision-Making on Surgery or Active Surveillance for Low-Risk Papillary Thyroid Cancer. Thyroid. 2020 Jul;30(7):999-1007. doi: 10.1089/thy.2019.0592. Epub 2020 Apr 8. PMID 32126932
- See also: Protocol manuscript - PMID: 29654030 — https://bmjopen.bmj.com/content/bmjopen/8/4/e020298.full.pdf
- See also: Study website — http://thyroidcancerstudy.ca